CLINICAL TRIAL: NCT04866563
Title: A Phase 2 Study to Assess the Efficacy and Safety of AX-8 in Patients With Chronic Cough
Brief Title: A Study of Efficacy and Safety of AX-8 in Chronic Cough
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axalbion SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AX8-003; 2021-000844-23 (EudraCT Number)
Record Dates: First submitted 2021-04-23; First posted 2021-04-30 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- AX-8 to Placebo, Part 1 of the study (Experimental): AX-8 BID, taken for 2 weeks, followed by a 1-week washout period and then Placebo BID, taken for 2 weeks.
  Interventions: Drug: AX-8, Part 1 of the study; Drug: Placebo, Part 1 of the study
- Placebo to AX-8, Part 1 of the study (Experimental): Placebo BID, taken for 2 weeks, followed by a 1-week washout period and then AX-8 BID, taken for 2 weeks.
  Interventions: Drug: AX-8, Part 1 of the study; Drug: Placebo, Part 1 of the study
- AX-8 to Placebo, Part 2 of the study (Experimental): AX-8 TID, taken for 2 weeks, followed by a 1-week washout period and then Placebo BID, taken for 2 weeks.
  Interventions: Drug: AX-8, Part 2 of the study; Drug: Placebo, Part 2 of the study
- Placebo to AX-8, Part 2 of the study (Experimental): Placebo TID, taken for 2 weeks, followed by a 1-week washout period and then AX-8 BID, taken for 2 weeks.
  Interventions: Drug: AX-8, Part 2 of the study; Drug: Placebo, Part 2 of the study

INTERVENTIONS:
Drug: AX-8, Part 1 of the study — orally disintegrating tablets, BID
  Arms: AX-8 to Placebo, Part 1 of the study; Placebo to AX-8, Part 1 of the study
Drug: Placebo, Part 1 of the study — orally disintegrating tablets, BID
  Arms: AX-8 to Placebo, Part 1 of the study; Placebo to AX-8, Part 1 of the study
Drug: AX-8, Part 2 of the study — orally disintegrating tablets, TID
  Arms: AX-8 to Placebo, Part 2 of the study; Placebo to AX-8, Part 2 of the study
Drug: Placebo, Part 2 of the study — orally disintegrating tablets, TID
  Arms: AX-8 to Placebo, Part 2 of the study; Placebo to AX-8, Part 2 of the study

SUMMARY:
This is a randomized, double-blind, placebo-controlled, crossover, multicenter study of AX-8 in participants with unexplained or refractory chronic cough designed to evaluate the effectiveness of AX-8 in reducing cough frequency.

ELIGIBILITY:
Inclusion Criteria:

* Chest radiograph or computed tomography (CT) of the thorax approximately 12 months before screening not demonstrating any abnormality considered to be significantly contributing to the chronic cough
* Have a diagnosis of refractory chronic cough (RCC) or unexplained chronic cough (UCC) for at least one year
* Women of childbearing potential and their male partners must use 2 acceptable methods of contraception
* Male subjects and their female partners of childbearing potential must use 2 acceptable methods of contraception
* Have provided written informed consent

Exclusion Criteria:

* Positive diagnostic nucleic acid test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)
* Current smoker (including e-cigarettes), individuals who have given up smoking within the past 12 months, or individuals with a smoking history of 20 pack-years
* Treatment with an ACE-inhibitor as the potential cause of a subject's cough or requiring treatment with an ACE-inhibitor during the study or within 12 weeks prior to the Baseline Visit
* History of upper or lower respiratory tract infection or recent significant change in pulmonary status within 4 weeks
* History of cystic fibrosis
* Positive test for any drug of abuse
* History of malignancy within 5 years prior to the Baseline Visit
* History of infection or known active infection with human immunodeficiency (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* History of hypersensitivity or intolerance to AX-8 or other TRPM8 agonists or any of the excipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Part 1 of the study: Change from Baseline in objective cough frequency in the 8 hours after the first dose of the day (i.e., Dose 1) on the 1st day of treatment of each study period | Baseline (i.e., Days -1 and 22) and the 1st day of treatment (i.e., Days 1 and 23) of each study period
  Assessment of number of coughs per hour to be evaluated using a digital recording device
Part 2 of the study: Change from Baseline in objective cough frequency in the 4 hours after the first dose of the day (i.e., Dose 1) on the 1st day of treatment of each study period | Baseline (i.e., Days -1 and 22) and the 1st day of treatment (i.e., Days 1 and 23) of each study period
  Assessment of number of coughs per hour to be evaluated using a digital recording device

SECONDARY OUTCOMES:
Change from Baseline in awake cough frequency | Baseline (i.e., Days -1 and 22), the 1st day of treatment (i.e., Days 1 and 23) and the 14th day of treatment (i.e., Days 14 and 36) of each study period
  Assessment of awake coughs per hour (average hourly cough frequency while the participant is awake based on sound recordings), to be evaluated using a digital recording device
Change from Baseline in Cough Severity Visual Analog Scale (VAS) score | Baseline (i.e., Days -1 and 22), the 1st day of treatment (i.e., Days 1 and 23) and the 14th day of treatment (i.e., Days 14 and 36) of each study period
  Cough Severity is determined through the use of a 100 mm visual analogue scale (VAS) (ranging between 0 for "no cough" and 100 for "worst cough").
Incidence (percent of participants) of treatment-emergent adverse events (TEAEs) | From first dose of study drug (i.e., Dose 1 on Day 1) to follow-up visit (i.e., Day 50, included)
  TEAEs are defined as those AEs (i.e., a new event or an exacerbation of a pre-existing condition) occurring on or after the first study dosing (i.e., Dose 1 on Day 1).
Incidence (percent of participants) of serious adverse events (SAEs) | From screening visit (i.e., Days -21 to -2) to follow-up visit (i.e., Day 50, included)
  An SAE is an adverse events occurring during any study phase and that fulfils one or more of the following: results in death, is life-threatening, requires patient hospitalization or results in prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a significant or important medical event, or is a congenital anomaly/birth defect in the offspring of a subject who received study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Axalbion Therapeutics, LTD.
Locations (16):
- United Kingdom (16):
  - Axalbion Study Site 4406, Birmingham, England
  - Axalbion Study Site 4404, Broughton, England
  - Axalbion Study Site 4409, Chelmsford, England
  - Axalbion Study Site 4413, Coventry, England
  - Axalbion Study Site 4401, London, England
  - Axalbion Study Site 4402, London, England
  - Axalbion Study Site 4410, London, England
  - Axalbion Study Site 4403, Manchester, England
  - Axalbion Study Site 4405, North Shields, England
  - Axalbion Study Site 4417, Orpington, England
  - Axalbion Study Site 4407, Oxford, England
  - Axalbion Study Site 4411, Preston, England
  - Axalbion Study Site 4412, Shipley, England
  - Axalbion Study Site 4408, Newport, Wales
  - Axalbion Study Site 4414, Belfast
  - Axalbion Study Site 4415, Northwood

IPD SHARING:
Plan to Share IPD: No